CLINICAL TRIAL: NCT04076410
Title: Efficacy of New Lenses in Abolishing Photoparoxysmal Responses in Paediatric Patients With Photosensitive Epilepsy (PSE)
Brief Title: Efficacy of Lenses in Abolishing Photoparoxysmal Responses
Acronym: PPRs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Collaborators: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ana Checa-Ros, MD, PhD, Honorary Research Fellow, Aston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 284-2019-CR; 266497 (Other: Health Research Authority, UK); 20/EM/0030 (Other: REC Reference Number)
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Reflex Epilepsy, Photosensitive; Eyeglasses
Keywords: photosensitivity; pattern sensitivity; Electroencephalography; Photic Stimulation; Pattern Stimulation; photoparoxysmal response; Light, Visible; Red Colour; Blue Light; children; epilepsy; standardized photoparoxysmal response range
MeSH Terms: conditions — Epilepsy, Reflex; Photosensitivity Disorders; Erythema; Epilepsy

STUDY DESIGN:
Intervention Model Description: Participants will be recruited among those patients (both males and females) from 5 to 18 years with suspected or confirmed diagnosis of generalised epilepsy with photosensitivity or photosensitive epilepsy (PSE) who comply with the established inclusion criteria.
  No control patients will be required, since each patient will be tested with the different lenses in a specific order and will be, in turn, his/her own control. No randomisation will be carried out in our study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5 Lenses (Experimental): The five lenses will be tested in each patient following always the same specific order, with the most protective lenses tested first (Z1).
  Z1F133 (Zeiss Clarlet Z1) is a CE marked device manufactured by Carl Zeiss Vision International GmBH (Aalen, Germany).
  Our lenses are CE marked devices manufactured by Cerium Optical Products (Kent, UK).
  Interventions: Device: Z1 lens; Device: Experimental Lens 1; Device: Experimental Lens 2; Device: Experimental Lens 3; Device: Experimental Lens 4

INTERVENTIONS:
Device: Z1 lens — CE marked device
  Other Names: Zeiss F133
Device: Experimental Lens 1 — CE marked device
Device: Experimental Lens 2 — CE marked device
Device: Experimental Lens 3 — CE marked device
Device: Experimental Lens 4 — CE marked device

SUMMARY:
Background. Blue lenses that filter out red light have been proposed as a new therapeutic alternative for patients with PSE, such as the lens Zeiss Clarlet Z1. This lens only allows a small overall quantity of visible light, and particularly a minimum percentage of red light, to pass through. However, these characteristics entail two main pitfalls: reduced applicability in high- latitude regions and lack of transmission for the red and yellow colors. The latter would mainly expose patients to the other colors that compose the visible light, and particularly to the blue visible light. This exposure might be damaging for their eyes in the long term, as it has been reported in some studies.

Aim. To determine whether four new lenses with different spectral characteristics are not inferior in efficacy to Z1 to reduce the PPRs in patients with PSE.

Participants. Patients between 5-18 years with suspected or confirmed PSE, referred to the Neurophysiology Service at Birmingham Children's Hospital (BCH) for an EEG with IPS/pattern stimulation.

Objectives & Outcomes:

1.A) Primary Objective: To evaluate the reduction/suppression produced by four new lenses in the PPRs shown by patients with PSE during an EEG with IPS/pattern stimulation, and compare it with the reduction provoked by the Z1 lens in the same individuals.

1. B) Primary Outcome: reduction/suppression in both the PPR and the standardized photoparoxysmal response range (SPR) for IPS and pattern stimulation.
2. A) Secondary Objectives:

   * To obtain feedback from the patients who acquire a pair of our lenses regarding tolerability, overall adherence to treatment and improvement in the quality of life.
   * Comparison of the reduction/suppression in the PPRs between our lenses and the Z1 lens in those retrospective patients with PSE seen between 2008-2017 at the Aston Brain Center.

2.B) Secondary Outcomes:

* Mean score obtained in adherence to treatment, tolerability, reduction in seizure frequency and autonomy according to the patient/parents or carers satisfaction questionnaires.
* Reduction/suppression in both the PPR and the standardized photoparoxysmal response range (SPR) for IPS and pattern stimulation in those patients recruited at the Aston Brain Center.

DETAILED DESCRIPTION:
1. BACKGROUND

   Photosensitive epilepsy (PSE) is the most common of reflex epilepsies and represents approximately 10% of all new cases of epilepsy in the age range 7-19 years (Harding & Jeavons, 1994). Photosensitivity is the nuclear feature of PSE, in which seizures are provoked by light stimuli or visual patterns, such as lines, gratings or checkerboards (Yalçin, Kaymaz, & Forta, 2000)(Fisher, Harding, Erba, Barkley, & Wilkins, 2005). Therefore, usual external triggers of seizures in the daily life of patients with PSE are sunlight and screens, like televisions (TVs), video games and computer displays. Photic/pattern sensitivity can be detected on the electroencephalogram (EEG) by the presence of a specific abnormality, called the 'photoparoxysmal response' (PPR), which is usually evoked by intermittent photic stimulation (IPS) or pattern stimulation, respectively (Quirk et al., 1995). Red color (wavelength around 600-700nm) has been proposed to be the most provocative stimulus among the primary colors to trigger photosensitivity/pattern-sensitivity in these patients (Fisher et al., 2005)(Guerrini & Genton, 2004).

   There are certain preventive measures to avoid triggering external stimuli which are particularly useful in PSE patients, but pharmacological treatment is required when seizures are not controlled by preventive measures or when photic or pattern-induced seizures coexist with spontaneous seizures. However, adverse effects of antiepileptic drugs (AEDs) and the relapse percentage after medication withdrawal, which may be nearly 50% (Verrotti et al., 2014), drove investigators to seek other therapeutic alternatives, such as the use of blue lenses that filter out red light. To date, the most extensively investigated lens has been Zeiss Clarlet Z1, which abolished PPRs in 75.9% of 610 patients (Giuseppe Capovilla et al., 2006). This effect was accounted for by the spectroscopic profile of Z1, that shows the minimal transmittance for the spectrum of red color (600-700 nm) (G Capovilla et al., 1999) and a luminous transmittance for the visible spectrum (τν) around 7%.

   However, Z1 transmittance characteristics have two main limitations for its use in everyday life: 1) it is a very dark lens and not practical in high-latitude regions, where the number of sunlight hours is reduced; 2) its lack of transmission in the red and yellow parts of the spectrum determines that people using Z1 are almost completely exposed to blue visible light, which has been associated with the appearance of ophthalmological diseases in the long term, such as age-related macular degeneration (AMD) ("blue-light hazard" phenomenon) (Mainster, 2006).
2. RATIONALE

   In light of these limitations, we hypothesized that a new type of lenses created by improving some spectral characteristics of Z1 could also be helpful for patients with PSE. This is the reason why we have designed four new lenses at the Aston Brain Center (ABC, Aston University) in collaboration with the Aston University Vision Sciences Department. These new lenses were firstly tested in those patients with PSE referred to the ABC between 2008-2017, when this center was the referral site in West Midlands to perform an EEG with photic/pattern stimulation.

   To date, no lens has demonstrated similar efficacy to Z1 with improved transmittance characteristics. Our new lenses may become an alternative or adjuvant therapy for paediatric and adult patients with PSE, leading to a reduction in the necessary dose of medication, with consequently less probability of adverse effects and an overall improvement in the quality of life.
3. AIM AND OBJECTIVES

The aim of our study is to demonstrate that our lenses are not inferior in efficacy to reduce the PPRs in comparison with Z1 in a sample of children and adolescents with PSE.

1. The primary objective of this study is to investigate the efficacy of these four lenses in suppressing the PPRs evoked by IPS and/or pattern stimulation in a sample of pediatric patients with PSE recruited at the Birmingham Women's and Children's NHS Foundation Trust (BWCH), and compare their results with those obtained with Z1 in the same patient.
2. Our secondary objectives are:

   * To collect the retrospective information (clinical and EEG data) of those PSE patients who were seen between 2008 and 2017 at the ABC, where the lenses were firstly tested before moving the equipment to the BWCH.
   * To obtain feedback from the patients who finally acquire a pair of our lenses in relation to the overall adherence to treatment, tolerability and improvement in the quality of life. To achieve this objective, we will send a patient satisfaction questionnaire (PSQ) to these patients approximately 6 months after purchasing the lenses.

     4. DESIGN

This is a single-arm clinical trial. We will carry out two types of study: a prospective (forward) study recruiting patients at BWCH and also a retrospective (backwards) study collecting those patients seen at the ABC between 2008 and 2017. In both studies, data analysis will take place at Aston University after being pseudonymized.

5. METHODS

5.1. Recruitment

Prospective study (BWCH, Aston University):

Patients (either males or females) from 5 to 18 years with suspected or confirmed diagnosis of generalised epilepsy with photosensitivity or photosensitive epilepsy (PSE) who are referred to the Neurophysiology Service at BCH for an EEG with IPS/pattern stimulation to confirm the diagnosis or check evolution, whether they are taking AEDs or not. Participants will be able to maintain concentration during the procedure, follow simple commands given by the NHS PI and have the capacity to assent (under 16 years) or consent (16-18 years) to participate after checking that they have understood the purpose of the study.

Retrospective study (Aston University):

•Selection criteria followed in the retrospective study conducted at the ABC were the same, except for the age criterion, since adult patients were also seen at the ABC.

5.2. Trial Procedures

Prospective study (BWCH, Aston University):

* On the first visit to the BWCH, a standardised procedure for EEG with IPS (Kasteleijn-Nolst Trenité et al., 2012) will be performed, followed by stimulation with visual patterns (stationary vertical grids at different spatial frequencies on a screen). If PPRs are shown in response to IPS/pattern stimulation, lenses will be tested to evaluate the relative reduction produced by our lenses & Z1 on the PPRs evoked by IPS/pattern testing. This reduction will be determined by the change in both the type of PPR and the standardized photoparoxysmal response range (SPR).
* If our lenses are effective and patients/families decide to acquire one of them, they will be asked to fill in a Likert-scale PSQ approximately 6 months after purchasing the lenses. This information will provide us with some feedback on the overall adherence to treatment, tolerability and improvement in the quality of life.

5.2.2) Retrospective study (Aston University): it will consist in the same procedures as the prospective study, but in this case the PSQ was not sent to patients/families.

6. DATA ANALYSIS

A minimum sample size of 76 patients was obtained based upon data collected from a previous pilot study, taking into consideration a power value of 80%, an alpha value of 5% and a non-inferiority margin of 0.03.

For each patient, we will compare the reduction/suppression on both the PPR and the SPR between the different lenses (α=0.05). PSQ results will be expressed by the percentages of patients/parents who marked a particular response in these multiple-choice questionnaires.

Missed data (patients who finally drop out of the study) will not be considered for analysis purposes.

7. ETHICAL CONSIDERATIONS

All procedures conducted will comply with the Declaration of Helsinki as revised in 2013, the Data Protection Act 1998 and Local Information Governance protocols. Consent will be sought from parents/legal guardians and patients over 15 years, as well as assent in the case of younger patients.

Only pseudonymized raw data will be available for sharing outside of the department as the analysis is to be performed by the PI-based at the sponsor site (Aston University). Data storage will be in keeping with the Trust Information Governance policies.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Children and adolescents between 5-18 years with suspected or confirmed diagnosis of photosensitive epilepsy (PSE), whether they are taking antiepileptic medication or not.
   2. Capacity to:

      * maintain concentration during the procedure
      * follow simple commands
      * assent (under 16 years) or consent (16-18 years) to participate after understanding the purpose of the study.
2. Exclusion Criteria:

   1. Presence of a condition that may compromise the ability to tolerate the procedure and/or the capacity to assent or consent, such as:

      * intellectual disability
      * attention-deficit/hyperactivity disorder
      * autism spectrum disorders
      * difficulties to understand verbal/written explanations in English
   2. Refusal to participate
   3. Generalized seizure during the EEG procedure.
   4. Female patients suspected or known to be pregnant.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
PPR change | Baseline (First visit T0)
  Relative change in the photoparoxysmal response grade
SPR change | Baseline (First visit T0)
  Relative change in the standardized photoparoxysmal response range (SPR)

SECONDARY OUTCOMES:
Adherence and tolerability to lenses in everyday life | 6 months after acquiring the lenses (T6)
  The score obtained in the different sections of the Patient Satisfaction Questionnaire [on a scale from 1 (worst outcome) to 5 (best outcome)]

CONTACTS AND LOCATIONS:
Overall Officials: Bryony Carr, BSc, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust; Ana Checa-Ros, MD, PhD, Principal Investigator — Aston University, Birmingham, UK; Sukhvir Wright, MD, PhD, Study Chair — Aston University
Locations (2):
- United Kingdom (2):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, West Midlands
  - Aston University, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No
All data recruited at BCH and at the ABC will be pseudonymized before being shared with the PI at Aston University to protect patient confidentiality.

REFERENCES:
- [Background] Capovilla G, Beccaria F, Romeo A, Veggiotti P, Canger R, Paladin F. Effectiveness of a particular blue lens on photoparoxysmal response in photosensitive epileptic patients. Ital J Neurol Sci. 1999 Jun;20(3):161-6. doi: 10.1007/s100720050026. PMID 10541598
- [Background] Capovilla G, Gambardella A, Rubboli G, Beccaria F, Montagnini A, Aguglia U, Canevini MP, Casellato S, Granata T, Paladin F, Romeo A, Stranci G, Tinuper P, Veggiotti P, Avanzini G, Tassinari CA. Suppressive efficacy by a commercially available blue lens on PPR in 610 photosensitive epilepsy patients. Epilepsia. 2006 Mar;47(3):529-33. doi: 10.1111/j.1528-1167.2006.00463.x. PMID 16529617
- [Background] Fisher RS, Harding G, Erba G, Barkley GL, Wilkins A; Epilepsy Foundation of America Working Group. Photic- and pattern-induced seizures: a review for the Epilepsy Foundation of America Working Group. Epilepsia. 2005 Sep;46(9):1426-41. doi: 10.1111/j.1528-1167.2005.31405.x. PMID 16146439
- [Background] Guerrini R, Genton P. Epileptic syndromes and visually induced seizures. Epilepsia. 2004;45 Suppl 1:14-8. doi: 10.1111/j.0013-9580.2004.451011.x. PMID 14706039
- [Background] Harding, G., & Jeavons, P. (1994). Photosensitive Epilepsy: Clinics in Developmental Medicine. London, UK: McKeith Press.
- [Background] Kasteleijn-Nolst Trenite D, Rubboli G, Hirsch E, Martins da Silva A, Seri S, Wilkins A, Parra J, Covanis A, Elia M, Capovilla G, Stephani U, Harding G. Methodology of photic stimulation revisited: updated European algorithm for visual stimulation in the EEG laboratory. Epilepsia. 2012 Jan;53(1):16-24. doi: 10.1111/j.1528-1167.2011.03319.x. Epub 2011 Nov 16. PMID 22091642
- [Background] Mainster MA. Violet and blue light blocking intraocular lenses: photoprotection versus photoreception. Br J Ophthalmol. 2006 Jun;90(6):784-92. doi: 10.1136/bjo.2005.086553. PMID 16714268
- [Background] Quirk JA, Fish DR, Smith SJ, Sander JW, Shorvon SD, Allen PJ. Incidence of photosensitive epilepsy: a prospective national study. Electroencephalogr Clin Neurophysiol. 1995 Oct;95(4):260-7. doi: 10.1016/0013-4694(95)00118-i. PMID 8529557
- [Background] Verrotti A, Grosso S, D'Egidio C, Parisi P, Spalice A, Pavone P, Capovilla G, Agostinelli S. Valproate in adolescents with photosensitive epilepsy with generalized tonic-clonic seizures only. Eur J Paediatr Neurol. 2014 Jan;18(1):13-8. doi: 10.1016/j.ejpn.2013.06.006. Epub 2013 Jul 26. PMID 23891468
- [Background] Yalcin AD, Kaymaz A, Forta H. Reflex occipital lobe epilepsy. Seizure. 2000 Sep;9(6):436-41. doi: 10.1053/seiz.2000.0424. PMID 10986003